CLINICAL TRIAL: NCT06744088
Title: Clinical Outcomes Of Modified Del Nido Cardioplegia In Adult And Pediatric Cardiac Surgery; A Multicentered Cross-Sectional Study
Brief Title: Clinical Outcomes Of Modified Del Nido Cardioplegia In Adult And Pediatric Cardiac Surgery
Status: Active, not recruiting | Type: Observational
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Other Study IDs: MSAHS/Batch-Spring23/007
Record Dates: First submitted 2024-12-17; First posted 2024-12-20 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Cardiac Events
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Del Nido cardioplegia solution

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Combination Product: Del Nido cardioplegia — To assess the clinical outcomes of modified Del Nido cardioplegia in cardiac surgeries across different age groups,

SUMMARY:
"Introduction: Modern cardiac surgery prioritizes myocardial protection, incorporating various strategies including cardioplegia to preserve heart function during surgery. The Del Nido (DN) cardioplegia solution, initially for pediatric use, shows promise in adult surgeries due to its longer protection duration and reduced re-dosing needs. However, its efficacy in adults remains under-researched.

DETAILED DESCRIPTION:
This study aims to evaluate the clinical outcomes of modified Del Nido cardioplegia in adult and pediatric cardiac surgeries, comparing intraoperative and postoperative metrics to provide evidence on its efficacy and safety.

To assess the clinical outcomes of modified Del Nido cardioplegia in cardiac surgeries across different age groups, focusing on myocardial protection, hemodynamic stability, surgical outcomes, recovery, and complications.

ELIGIBILITY:
Inclusion Criteria:

* All Pediatric patients with congenital heart diseases.
* Individuals who are capable of giving their informed permission;
* Stable patients undergoing surgical procedures that involve cardiopulmonary bypass and cardiac arrest;
* isolated CABG surgery, or simultaneous CABG;
* isolated single-valve surgery or multiple value procedures.

Exclusion Criteria:

* Previous cardiac surgery
* Patients with preoperative inotropic pharmacologic support
* Patients receiving preoperative mechanical circulatory support,
* Patients with an implanted pacemaker or implantable cardioverter-defibrillator,
* Patients undergoing cardiac surgical procedures
* Patients who underwent off-pump or beating heart CABGs
* Ventilation for the night was scheduled because of severe pulmonary arterial hypertension.
* mediastinal drain causing a delay in extubation, or the need to reopen for bleeding or tamponade.

Ages: 1 Year to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Modern cardiac surgery prioritizes myocardial protection, incorporating various strategies including cardioplegia to preserve heart function during surgery. The Del Nido (DN) cardioplegia solution, initially for pediatric use, shows promise in adult surgeries due to its longer protection duration and reduced re-dosing needs.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2024-02-28 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
the Bypass time | up to 12 Months
postoperative mortality | 12 Months

CONTACTS AND LOCATIONS:
Locations (1):
- Peshawar, Peshawar, Khyber Pakhtunkhwa, Pakistan

IPD SHARING:
Plan to Share IPD: No